CLINICAL TRIAL: NCT04319796
Title: European Registry on Rare Neurological Diseases
Acronym: ERN-RND reg
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Prof. Dr. Ludger Schöls, Clinical Professor, University Hospital Tuebingen
Other Study IDs: ERN-RND registry
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Rare Diseases
Keywords: Rare Diseases; Ataxia; Hereditary Spastic Spinal Paralysis; Neurodegeneration with Brain Iron Accumulation; Leukodystrophy; Dystonia; Atypical Parkinsonism; Huntington's Disease; Chorea Huntington; European Reference Network on Rare Neurological Diseases; Frontotemporal Dementia
MeSH Terms: conditions — Rare Diseases; Ataxia; Pantothenate Kinase-Associated Neurodegeneration; Dystonia; Huntington Disease; Chorea; Frontotemporal Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 25 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Ataxia & HSP: Patients suffering of Ataxia or HSP or probands who are at risk to develop such a disease since they are first degree relatives of patients affected by these Rare Neurological Disease (RND).
  Interventions: Other: Data set as defined by the ERN Research Workgroup of the European Commission
- Leukodystrophies: Patients suffering of Leukodystrophies or probands who are at risk to develop such a disease since they are first degree relatives of patients affected by this RND.
  Interventions: Other: Data set as defined by the ERN Research Workgroup of the European Commission
- Frontotemporal Dementia: Patients suffering of Frontotemporal Dementia or probands who are at risk to develop such a disease since they are first degree relatives of patients affected by this RND.
  Interventions: Other: Data set as defined by the ERN Research Workgroup of the European Commission
- Dystonia, Paroxysmal Disorders and Neurodegeneration with: Patients suffering of Dystonia, Paroxysmal Disorders and Neurodegeneration with Brain Iron Accumulation (NBIA) or probands who are at risk to develop such a disease since they are first degree relatives of patients affected by these RND.
  Interventions: Other: Data set as defined by the ERN Research Workgroup of the European Commission
- Atypical Parkinsonism: Patients suffering of Atypical Parkinsonism or probands who are at risk to develop such a disease since they are first degree relatives of patients affected by this RND.
  Interventions: Other: Data set as defined by the ERN Research Workgroup of the European Commission
- Huntington's Disease & Choreas: Patients suffering of Huntington's Disease or Choreas or probands who are at risk to develop such a disease since they are first degree relatives of patients affected by these RND.
  Interventions: Other: Data set as defined by the ERN Research Workgroup of the European Commission

INTERVENTIONS:
Other: Data set as defined by the ERN Research Workgroup of the European Commission — The ERN-RND registry will be restricted to the minimum data set as defined by the ERN Research Workgroup of the European Commission. This includes the following data:
  * Name of specialist center
  * Pseudonym:
  * Date of birth: For confidentiality reasons the ERN-RND registry will restrict this information to the Year of birth
  * Sex
  * Date of death: For confidentiality reasons the ERN-RND registry will restrict this information to the Year of death
  * Age of onset
  * Orphacode for specific rare disease: https://www.orpha.net/consor/cgi-bin/Disease_Search.php?lng=DE
  * Online Mendelian Inheritance in Man (OMIM) code as defined for genetic diseases: https://www.omim.org/
  * Human Phenotype Ontology (HPO) terms for key features: https://hpo.jax.org/app/
  * Agreement to be contacted for research purposes: Yes/No
  * Biological samples (Yes / No)
  * Link to a biobank (Link / No)
  * Classification of disability (Disease group specific score)

SUMMARY:
The recent implementation of European Reference Networks for Rare Diseases (ERNs) is an unprecedented move to improve the care of patients suffering from rare health disorders by transnational collaboration. ERN-RND, the ERN for Rare Neurological Diseases, oversees more than 35,000 patients in 31 specialist centers in 13 countries. The ERN-RND registry aims to gather information on patient cohorts in the multiple specialist centers and to provide an overview on patient numbers principally accessible for translational studies.

DETAILED DESCRIPTION:
The ERN-RND (European Reference Network on Rare Neurological Diseases) Registry aims to establish a demographic platform for collection of relevant core patient information. This will be accomplished by the construction and implementation of a single data base encompassing all rare neurological diseases in pediatric and adult patients (the ERN-RND Registry), which will collect information according to the "Set of common data elements for Rare Diseases Registration" as it has been defined by the European Commission.

The ERN-RND network covers the following six disease groups in patients of all age groups: (i) Ataxia and Hereditary Spastic Spinal Paralysis (HSP), (ii) Leukodystrophies, (iii) Frontotemporal Dementia, (iv) Dystonia, Paroxysmal Disorders and Neurodegeneration with Brain Iron Accumulation (NBIA), (v) Atypical Parkinsonism and (vi) Huntington's Disease & Choreas.

ELIGIBILITY:
Inclusion Criteria:

Patients suffering of one of the rare neurological diseases indicated below or probands who are at risk to develop such a disease since they are first degree relatives of patients affected by a RND including:

* Ataxia and HSP
* Leukodystrophies
* Frontotemporal Dementia
* Dystonia, Paroxysmal Disorders and Neurodegeneration with Brain Iron Accumulation (NBIA)
* Atypical Parkinsonism
* Huntington's Disease & Choreas

Exclusion Criteria:

• Missing informed consent of the patient and/ or their parents

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients suffering of one of the rare neurological diseases indicated according to the inclusion criteria or probands who are at risk to develop such a disease since they are first degree relatives of patients affected by a RND. Patients visiting in Tübingen, Germany the specialist center Department of Neurology and/ or the Department of Neuropediatric Diseases at the University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Representative cohorts of RND patients | Day 1
  The register study aims to compile representative cohorts of RND patients and provide demographic data for the planning of translational studies. As all of the index diseases are rare the primary goal is to reach as large cohorts as possible.

CONTACTS AND LOCATIONS:
Overall Officials: Ludger Schöls, Prof. Dr., Study Director — University Hospital Tübingen

IPD SHARING:
Plan to Share IPD: Yes
The full pseudonymised dataset will be exported once a year as an Excel file that is made accessible in an encrypted form to the coordinators of each specialist center who contribute to the ERN-RND registry. To this end the encrypted dataset will be provided in a specific folder of the Hertie Institute for Clinical Brain Research Tübingen, Germany (HIH) cloud for a limited amount of time (one week). Coordinators of all ERN-RND health care providers will get access to this folder to download the encrypted file. In addition, they will receive a password that enables decryption of the file. Each coordinator needs to confirm a priori with its local institutional review board the issues of data storage. This is part of the local project plan, patient information and consent that is premise for data entry. This procedure enables each center who contributes data to consider studies of their special interest within the ERN.
Supporting Information: Analytic Code
Time Frame: Data will become available after analysis and unlimited.
Access Criteria: Authorized users within the participating organizations.